CLINICAL TRIAL: NCT04573881
Title: The HistoSonics System for Treatment of Primary and Metastatic Liver Tumors Using Histotripsy (#HOPE4LIVER EU/UK)
Acronym: #HOPE4LIVER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP1473
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Liver Neoplasms; Hepatocellular Carcinoma; Liver Metastases
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: This trial is a single arm, non-randomized, multicenter, prospective trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HistoSonics System (Experimental)
  Interventions: Device: HistoSonics System

INTERVENTIONS:
Device: HistoSonics System — The HistoSonics System - intended for the destruction of liver tissue using histotripsy, a non-thermal, mechanical process using focused ultrasound.
  Other Names: Histotripsy

SUMMARY:
This trial is a single arm, non-randomized prospective trial. The objective of this trial is to evaluate the efficacy and safety of the HistoSonics System for the treatment of primary or metastatic tumors located in the liver.

DETAILED DESCRIPTION:
This trial is a single arm, non-randomized, multicenter, prospective trial. Following histotripsy treatment of liver tumor(s), subjects will undergo imaging ≤36 hours post-index procedure to determine technical success. Subjects will then be followed for 30 days. Additionally, subjects will be evaluated at 6 months and followed annually for up to five (5) years post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subject has signed the Ethics Committee (EC) or Institutional Review Board (IRB) approved trial Informed Consent Form (ICF) prior to any trial related tests/procedures and is willing to comply with trial procedures and required follow-up assessments
3. Subject is diagnosed with hepatocellular carcinoma (HCC) or liver metastases (mets) from other primary cancers

   * Subject that is an HCC patient must have a targetable lesion(s) which meets the United Network for Organ Sharing and Organ Procurement and Transplantation Network (UNOS-OPTN) class 5 diagnostic criteria for HCC
   * Subject that is diagnosed with liver metastases must have prior diagnosis of primary tumor or metastatic tumor to identify the primary cancer type. Subjects must have untreated new or growing liver tumor(s) radiologically consistent with metastases. Note: A biopsy is required to confirm metastatic disease and the pathological results must be obtained prior to the index procedure (does not need to be a targeted tumor(s))
4. Subject is able to undergo general anesthesia
5. Subject has a Child-Pugh Score of A or B (up to B8)
6. Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) grade 0-2 at baseline screening
7. Subject meets the following functional criteria, ≤7 days prior to the planned index-procedure date:

   * Liver function: Alanine transaminase (ALT) <2.5x upper limit of normal (ULN) and Aspartate transaminase (AST) <2.5x ULN and bilirubin <2.5 ULN, and
   * Renal function: serum creatinine <2x ULN, and
   * Hematologic function: neutrophil count >1.0 x 10^9/L and platelet >50 x 10^9/L
8. Subject has an International Normalized Ratio (INR) score of <2.0 , ≤7 days prior to the planned index procedure date
9. Subject has not responded to and/or has relapsed and/or is intolerant of other available therapies including locoregional therapies, chemotherapy, immunotherapy and targeted therapies.
10. The tumor(s) selected for histotripsy treatment must be ≤3 cm in longest diameter
11. Subject has an adequate acoustic window to visualize targeted tumor(s) using ultrasound imaging
12. Subject has a maximum of three (3) tumors to be treated with histotripsy during the index procedure, regardless of how many tumors the subject has.

Note: If the subject is treated with surgical resection prior to the index procedure, the resection must be performed ≥2 weeks prior to the planned index-procedure date

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant or nursing (lactating) during the trial period
2. Subject is enrolled in another investigational trial and/or is taking investigational medication and/or has been treated with an investigational device ≤30-days prior to planned index procedure date
3. In the Investigator's opinion, the subject has co-morbid disease(s) or condition(s) that would cause undue risk and preclude safe use of the HistoSonics System
4. Subject has a serum creatinine >2.0 mg/dL or estimated glomerular filtration rate (EGFR) <30, unless on dialysis
5. Subject has major surgical procedure or significant traumatic injury ≤2 weeks prior to the planned index procedure or not fully recovered (CTCAE grade 1 or better) from side effects/complications of such procedure or trauma
6. Subject has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better from any adverse effects (except alopecia, fatigue, nausea, vomiting and peripheral neuropathy) related to previous anti-cancer therapy
7. Subject has a history of, or suspected to have, bleeding disorders that are uncorrectable
8. Subject has a coagulopathy that is uncorrectable
9. Subject has a planned cancer treatment (e.g. resection, chemotherapy, etc.) after the planned index-procedure date and prior to completion of the 30-day follow-up visit
10. Subject has previous treatment with bevacizumab that has not been discontinued >40 days prior to the planned index-procedure date
11. Subject has planned bevacizumab treatment prior to completion of the 30-day follow-up visit
12. Subject has previous treatments with chemotherapy and/or radiotherapy that has not been discontinued ≥2 weeks prior to the planned index-procedure date and has not recovered (CTCAE grade 1 or better) from related toxicity (except alopecia and peripheral neuropathy)
13. Subject has previous treatment with immunotherapies that has not been discontinued ≥4 weeks prior to the planned index-procedure date and has not recovered from related toxicity (CTCAE grade 1 or better)
14. Subject has a life expectancy less than six (<6) months
15. In the opinion of the Investigator, histotripsy is not a treatment option for the subject
16. Subject has a concurrent condition that, in the investigator's opinion, could jeopardize the safety of the subject or compliance with the protocol
17. Subjects' tumor(s) is not treatable by the System's working ranges (refer to User Manual)
18. Subject has a known sensitivity to contrast media and cannot be adequately pre-medicated
19. Subjects' targeted tumor(s) has/have had prior locoregional therapy (e.g. ablation, embolization, radiation)
20. Subject is eligible for surgical resection
21. Targeted tumor(s) treatment volume overlaps a non-targeted tumor visible via imaging
22. The targeted tumor(s) is not clearly visible with diagnostic ultrasound and computed tomography (CT) or magnetic resonance (MR) imaging
23. The targeted tumor(s) is located in liver segment 1
24. The Planned Treatment Volume intended to cover the targeted tumor includes or encompasses any portion of the main portal vein, common hepatic duct, common bile duct, gallbladder or stomach/bowel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2027-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi A Solbiati, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (6):
- Germany (2):
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitätsklinikum Magdeburg Klinik für Radiologie und Nuklearmedizin, Magdeburg
- Istituto Clinico Humanitas - Humanitas Mirasole S.P.A., Milan, Italy
- Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wah TM, Pech M, Thormann M, Serres X, Littler P, Stenberg B, Lenton J, Smith J, Wiggermann P, Planert M, Vidal-Jove J, Torzilli G, Solbiati L. A Multi-centre, Single Arm, Non-randomized, Prospective European Trial to Evaluate the Safety and Efficacy of the HistoSonics System in the Treatment of Primary and Metastatic Liver Cancers (#HOPE4LIVER). Cardiovasc Intervent Radiol. 2023 Feb;46(2):259-267. doi: 10.1007/s00270-022-03309-6. Epub 2022 Nov 15. PMID 36380155
- [Result] Mendiratta-Lala M, Wiggermann P, Pech M, Serres-Creixams X, White SB, Davis C, Ahmed O, Parikh ND, Planert M, Thormann M, Xu Z, Collins Z, Narayanan G, Torzilli G, Cho C, Littler P, Wah TM, Solbiati L, Ziemlewicz TJ. The #HOPE4LIVER Single-Arm Pivotal Trial for Histotripsy of Primary and Metastatic Liver Tumors. Radiology. 2024 Sep;312(3):e233051. doi: 10.1148/radiol.233051. PMID 39225612
- [Result] Ziemlewicz TJ, Critchfield JJ, Mendiratta-Lala M, Wiggermann P, Pech M, Serres-Creixams X, Lubner M, Wah TM, Littler P, Davis CR, Narayanan G, White SB, Ahmed O, Collins ZS, Parikh ND, Planert M, Thormann M, Torzilli G, Solbiati LA, Cho CS. The #HOPE4LIVER Single-arm Pivotal Trial for Histotripsy of Primary and Metastatic Liver Tumors: One-year Update of Clinical Outcomes. Ann Surg. 2025 Dec 1;282(6):908-916. doi: 10.1097/SLA.0000000000006720. Epub 2025 Apr 9. PMID 40201962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was designed to enroll up to 45 participants; however, enrollment was stopped after 24 participants were enrolled due to completion of the primary analysis of #HOPE4LIVER US (NCT04572633). The primary analysis assessed the primary and secondary endpoints at 30 days using pooled data from #HOPE4LIVER EU/UK and #HOPE4LIVER US after a total of 40 evaluable participants enrolled between the two trials. Follow-up beyond 30 days is ongoing.
Period: Overall Study
Arm/Group | HistoSonics System
Started | 24
Completed | 0 (No participant completed the trial at 30 days. Primary outcomes were analyzed at 30 days. Follow up is ongoing.)
Not Completed | 24
Not completed — Participant in active follow-up at 30 days | 24

BASELINE CHARACTERISTICS:
Arm/Group | HistoSonics System
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  Other | 1
Type of tumor [Count of Participants; unit: Participants]
  Hepatocellular carcinoma | 7
  Liver metastasis | 17

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: Technical Success
Description: Technical success, defined as the treatment volume/treatment dimensions being greater than or equal to the targeted tumor, and with complete tumor coverage, via computed tomography (CT) or magnetic resonance (MR) imaging. [Core Laboratory Adjudicated]
Time Frame: ≤36 hours post-index procedure
Population: Four tumors had insufficient imaging data for the core laboratory to evaluate technical success.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: tumors
Arm/Group | HistoSonics System
Number analyzed (Participants) | 21
Number analyzed (tumors) | 22
percentage of tumors | 100 [100 to 100]

2. Primary Outcome: Primary Safety: Procedure-Related Major Complications
Description: Number of index procedure related major complications, including device-related events defined as Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher toxicities observed up to 30-days post index-procedure. [Clinical Events Committee Adjudicated]
Time Frame: 30 days post-index procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HistoSonics System
Number analyzed (Participants) | 24
percentage of participants | 12.5 [4.3 to 31.0]

3. Secondary Outcome: Secondary Efficacy: Technique Efficacy
Description: Technique efficacy, defined as the lack of a nodular or mass-like area of enhancement within or along the edge of the treatment volume assessed via CT or MR imaging at 30-days post-procedure. [Core Laboratory Adjudicated]
Time Frame: 30 days post-index procedure
Population: Five of the 22 tumors analyzed for technical success had missing or insufficient imaging data for the core laboratory to evaluate technique efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: tumors
Arm/Group | HistoSonics System
Number analyzed (Participants) | 17
Number analyzed (tumors) | 17
percentage of tumors | 100 [100 to 100]

4. Secondary Outcome: Secondary Safety: All Adverse Events
Description: Number of adverse events (serious and non-serious) reported within 30 days post-index procedure. [Clinical Events Committee Adjudicated]
Time Frame: 30 days post-index procedure
Measure: Number; unit: adverse events
Arm/Group | HistoSonics System
Number analyzed (Participants) | 24
adverse events | 38

ADVERSE EVENTS:
Time Frame: Enrollment through 30 days
Description: All adverse events were reported starting at the time the participant was enrolled in the trial to the 1-year visit interval or trial exit (whichever comes first). Data collection for adverse events is still ongoing.
Arm/Group | HistoSonics System
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HistoSonics System (N=24)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1)
Melaena/Melena (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HistoSonics System (N=24)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 4 (5)
Procedural pain (Injury, poisoning and procedural complications) | 6 (6)
Anaemia/Anemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (2)
Discomfort (General disorders) | 1 (1)
Localized oedema (General disorders) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hepatic hypoperfusion (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to completion of the primary analysis in #HOPE4LIVER US (NCT04572633) that included powered efficacy and safety hypothesis testing on combined US and EU/UK participants, #HOPE4LIVER EU/UK trial enrollment was stopped early. Therefore, there is an insufficient number of target participants needed to achieve target power and statistically reliable results for the primary endpoints for #HOPE4LIVER EU/UK.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04573881/Prot_SAP_000.pdf